CLINICAL TRIAL: NCT01037452
Title: A Phase II, Randomized, Double-blind, Placebo-controlled, Parallel Group Proof-of-Concept Trial to Assess Relief of Meal Induced Heartburn by a Combination of Lansoprazole 15 mg and Antacid Versus Lansoprazole 15 mg and Antacid (Calcium Carbonate and Magnesium Hydroxide) Alone
Brief Title: Proof of Concept Study Efficacy of an Antacid/Lansoprazole Combination for Relief of Heartburn
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Head, New Therapeutic Opportunities, Novartis
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 145-G-201
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Results first posted 2011-03-28 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Heartburn
Keywords: Heartburn; antacid; PPI; Lansoprazole; calcium carbonate; magnesium hydroxide; Relief of heartburn following ingestion of a heartburn-inducing meal
MeSH Terms: conditions — Heartburn | interventions — Calcium Carbonate; Magnesium Hydroxide; Lansoprazole; dihydroxyaluminum sodium carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- Combination product (Experimental): Calcium carbonate/magnesium hydroxide/Lansoprazole 15 mg tablet
  Interventions: Drug: Calcium carbonate/magnesium hydroxide/Lansoprazole 15 mg
- PPI alone (Active Comparator): Lansoprazole
  Interventions: Drug: Lansoprazole
- Antacid alone (Active Comparator): Calcium carbonate/magnesium hydroxide
  Interventions: Drug: Calcium carbonate/magnesium hydroxide
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcium carbonate/magnesium hydroxide/Lansoprazole 15 mg — Tablet
  Arms: Combination product
Drug: Lansoprazole — Tablet
  Arms: PPI alone
Drug: Calcium carbonate/magnesium hydroxide — Tablet
  Arms: Antacid alone
Drug: Placebo — Tablet
  Arms: Placebo

SUMMARY:
This study will investigate the safety and efficacy of an antacid/Lansoprazole combination product for the relief of heartburn after consuming a heartburn-inducing meal.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing heartburn in the past month if untreated
* Having heartburn that responds to heartburn medication
* Be willing to discontinue the use of heartburn treatment for 7 days prior to inclusion in the study.

Exclusion Criteria:

* Having history of erosive esophagitis or gastroesophageal reflux disease (GERD) diagnosed by a physician and confirmed by testing (endoscopy)
* Be unwilling to take only the study medication, and antacid provided as a rescue medication for relief of acute heartburn during the study.

"Other protocol-defined inclusion/exclusion criteria may apply"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-12; Primary Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis ., Study Director — Novartis
Locations (1):
- Anaheim, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination Product: Calcium carbonate/magnesium hydroxide/Lansoprazole 15 mg tablet, single dose
- PPI Alone: Lansoprazole 15 mg, single dose
- Antacid Alone: Calcium carbonate/magnesium hydroxide, single dose
- Placebo: Placebo, single dose
Period: Overall Study
Arm/Group | Combination Product | PPI Alone | Antacid Alone | Placebo
Started | 30 | 30 | 30 | 30
Completed | 30 | 30 | 30 | 30
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Product | PPI Alone | Antacid Alone | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 30 | 29 | 119
  >=65 years | 0 | 0 | 0 | 1 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 33.7 (11.5) | 30.4 (11.1) | 30.9 (13.3) | 31.9 (12.6) | 31.7 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 11 | 17 | 57
  Male | 15 | 16 | 19 | 13 | 63
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 30 | 30 | 120

OUTCOME MEASURES:

1. Primary Outcome: Measure: Number of Participants With no Heartburn (Post Treatment) Following Consumption of Heartburn-inducing Meal
Description: Participant reported severity of heartburn using a Visual Analog Scale (VAS)directly on CRF every 15 minutes until no heartburn reported or up to 5 hours after 1st heartburn-inducing meal, whichever occurred first. At this point in time, a diary was provided to participants to record any changes in severity of heartburn for 28 hours post treatment.
Time Frame: 1 day
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Combination Product | PPI Alone | Antacid Alone | Placebo
Number analyzed (Participants) | 30 | 30 | 30 | 30
participants | 0 [0.0 to 11.6] | 2 [0.8 to 22.1] | 1 [0.1 to 17.2] | 0 [0.0 to 11.6]

2. Secondary Outcome: Measure: Maximum Heartburn Intensity for Those Participants Who Experience Any Heartburn After the Heartburn-inducing Meals
Description: Heartburn severity was measured using a Visual Analog Scale, which was 100 milliimeters long.
  0 millimeters: None (no heartburn) 100 millimeters: Most severe
Time Frame: 1 day
Measure: Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Combination Product | PPI Alone | Antacid Alone | Placebo
Number analyzed (Participants) | 30 | 30 | 30 | 30
millimeters | 69.3 [62.8 to 75.8] | 61.2 [51.6 to 70.7] | 59.1 [50.5 to 67.8] | 56.9 [50.4 to 63.4]

3. Secondary Outcome: Measure: Maximum Heartburn Intensity for Those Participants Who Experience Any Nighttime Heartburn
Description: as for outcome 2
Time Frame: 1 day
Measure: Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Combination Product | PPI Alone | Antacid Alone | Placebo
Number analyzed (Participants) | 30 | 30 | 30 | 30
millimeters | 8.2 [0.4 to 16.0] | 7.0 [-1.0 to 15.0] | 4.7 [-0.9 to 10.2] | 4.0 [-1.6 to 9.6]

4. Secondary Outcome: Measure: Number of Participants That Reported an Adverse Event for the Combination Product, PPI Alone, Antacid Alone and Placebo.
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | Combination Product | PPI Alone | Antacid Alone | Placebo
Number analyzed (Participants) | 30 | 30 | 30 | 30
participants | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Combination Product | PPI Alone | Antacid Alone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less